CLINICAL TRIAL: NCT00788931
Title: A Phase Ib, Open-label, Two Arm Study of i.v. and Oral Panobinostat (LBH589) in Combination With i.v. Trastuzumab (Herceptin®) and i.v. Paclitaxel as Treatment for Adult Female Patients With HER2 Overexpressing Metastatic Breast Cancer (MBC)
Brief Title: A Trial l of Panobinostat Given in Combination With Trastuzumab and Paclitaxel in Adult Female Patients With HER2 Positive Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589C2114; 2007-004788-23 (EudraCT Number)
Record Dates: First submitted 2008-10-24; First posted 2008-11-11 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2012-11

CONDITIONS: HER-2 Positive Breast Cancer; Metastatic Breast Cancer
Keywords: Breast Cancer; HER2 positive; adult-female; LBH589; HDAC inhibitor; panobinostat; metastatic breast; adult female patients
MeSH Terms: conditions — Breast Neoplasms | interventions — Panobinostat; Trastuzumab; Paclitaxel

ARMS (2):
- IV LBH589 + trastuzumab + paclitaxel (Experimental): i.v. panobinostat
  Interventions: Drug: IV LBH589; Drug: trastuzumab; Drug: paclitaxel
- Oral LBH589 + trastuzumab + paclitaxel (Experimental): oral panobinostat
  Interventions: Drug: IV LBH589; Drug: Oral LBH589; Drug: trastuzumab; Drug: paclitaxel

INTERVENTIONS:
Drug: IV LBH589
Drug: Oral LBH589
  Arms: Oral LBH589 + trastuzumab + paclitaxel
Drug: trastuzumab
Drug: paclitaxel

SUMMARY:
The primary purpose of this study is to identify the maximum tolerated dose (MTD) of both intravenous and oral panobinostat when given in combination with trastuzumab and paclitaxel. The study will evaluate safety and efficacy of the combination in adult female patients with HER2+ metastatic breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 year old
* Confirmed HER2+ metastatic breast cancer
* Prior treatment and progression on trastuzumab
* Patients must have adequate organ functions
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1

Exclusion Criteria:

* Patients who have had surgery within last 2 weeks prior to starting the treatment
* Patients who receive concurrent therapy for brain metastases
* Impaired heart function or clinically significant heart disease
* Ongoing diarrhea
* Liver or renal disease with impaired hepatic or renal functions
* Concomitant use of any anti-cancer therapy or certain drugs
* Female patients who are pregnant or breast feeding
* Patients not willing to use an effective method of birth control Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-12; Primary Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose of oral panobinostat in combination with trastuzumab and paclitaxel. Determine the maximum tolerated dose of iv LBH in combination with trastuzumab and paclitaxel. | At least 21 day cycle for both arms

SECONDARY OUTCOMES:
Safety and tolerability throughout the study for both IV and oral arms to determine the recommended dose for phase ll trials. | 4 weeks after end of treatment
To evaluate the efficacy in the expansion phase of the trial when the MTD is defined. | throughout the study and 4 weeks after end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- Novartis Investigative Site, Mobile, Alabama, United States
- Novartis Investigative Site, Woodville, South Australia, Australia
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Liège
- Italy (2):
  - Novartis Investigative Site, Macerata, MC
  - Novartis Investigative Site, Aviano, PN
- Novartis Investigative Site, Amsterdam, Netherlands

REFERENCES:
- See also: Results for LBH589C2114 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=4342